CLINICAL TRIAL: NCT01423539
Title: A Phase II, Multicenter, Randomized, Controlled, Open-Label Study of Bendamustine + Rituximab With or Without Navitoclax in Patients With Relapsed Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Navitoclax in Addition to Bendamustine and Rituximab in Patients With Relapsed Diffuse Large B-Cell Lymphoma (NAVIGATE)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The NAVIGATE study has been terminated due to non-safety related reasons.
Sponsor: Genentech, Inc. (Industry)
Collaborators: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP27814
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; navitoclax; Rituximab

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: bendamustine; Drug: rituximab
- B (Experimental)
  Interventions: Drug: bendamustine; Drug: navitoclax; Drug: rituximab

INTERVENTIONS:
Drug: bendamustine — Intravenous repeating dose\n
Drug: navitoclax — Oral repeating dose\n
  Arms: B
Drug: rituximab — Intravenous repeating dose\n

SUMMARY:
This randomized, open-label, multicenter study will evaluate the efficacy and safety of navitoclax in addition to bendamustine and rituximab in patients with relapsed diffuse large B-cell lymphoma. Patients will be randomized to receive navitoclax in addition to bendamustine and rituximab or bendamustine and rituximab alone for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of diffuse large B-cell lymphoma
* Patients must have relapsed or developed progressive disease following salvage therapy, or must have relapsed or progressed following initial therapy and in the opinion of the investigator are medically unfit to receive high dose chemotherapy with autologous stem cell transplant (SCT) or other salvage therapy of higher priority
* Eastern cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients who have undergone STC must be more than 100 days from autologous stem cell infusion prior to first dose of study drug, must have recovered from any transplant related toxicity and must have adequate bone marrow function as defined by protocol independent of any growth factor support
* Patients who have not undergone SCT must have adequate bone marrow function as defined by protocol independent of any growth factor support
* Adequate coagulation, renal and hepatic function

Exclusion Criteria:

* Refractory DLBCL
* History of other malignancies within 2 years prior to initiation of study treatment except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin carcinoma, low-grade localized prostate cancer treated surgically with curative intent or one that carries a good prognosis, in situ ductal carcinoma of the breast treated with lumpectomy (with and without radiation) with curative intent
* Active infection requiring parenteral antibiotics or antiviral or antifungal agents
* Inherited or acquired bleeding diathesis, anticoagulant drugs or drugs that inhibit platelet function, underlying conditions that predisposes to abnormal bleeding, or refractoriness to platelet transfusions
* Clinically significant cardiovascular disease, New York Heart Association Grade II or greater congestive heart failure, or ventricular tachyarrhythmias requiring medication within 1 year prior to the initiation of study treatment
* Positive for hepatitis B, hepatitis C or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (time from randomization to progression, relapse or death of any cause) | up to approximately 33 months

SECONDARY OUTCOMES:
Clinical response rates (complete response/partial response/stable disease) | approximately 33 months
Duration of response | approximately 33 months
Overall survival | approximately 33 months
Safety: Incidence of adverse events | approximately 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (13):
- United States (13):
  - Fountain Valley, California
  - Hudson, Florida
  - Lawrenceville, Georgia
  - Centralia, Illinois
  - Harvey, Illinois
  - Terre Haute, Indiana
  - Hazard, Kentucky
  - Paducah, Kentucky
  - Rockville, Maryland
  - Jefferson City, Missouri
  - Great Falls, Montana
  - Newark, Ohio
  - Nashville, Tennessee